CLINICAL TRIAL: NCT02530450
Title: iPro Continuous Glucose Monitor in Children With Poorly Controlled Diabetes: A 6-Month, Randomized, Interventional Pilot Study
Brief Title: Continuous Glucose Monitor in Children With Poorly Controlled Diabetes
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: HSC20110049H
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: children; poor adherence; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Initially blinded to continuous glucose monitoring (CGM) data after 1st use Not blinded to continuous glucose monitoring data after 2nd and 3rd use
  Interventions: Device: continuous glucose monitoring (CGM)
- Group 2: Never blinded to continuous glucose monitoring (CGM) data
  Interventions: Device: continuous glucose monitoring (CGM)

INTERVENTIONS:
Device: continuous glucose monitoring (CGM) — All subjects in Groups 1 and 2 wore the CGM device at time points 0, 3 months, and 6 months. Group 1 did not review CGM data at time 0, but did review CGM data at time point 3 months and 6 months. Group 2 reviewed CGM data at all time points.
  Other Names: iPRO

SUMMARY:
The purpose of this study is to determine if the use of continuous glucose monitoring in a practical outpatient clinic setting in children with poorly controlled diabetes will lead to improved blood sugar control.

DETAILED DESCRIPTION:
The trial was designed as a six month, randomized, prospective, interventional pilot study of children with uncontrolled (HgbA1c > 8.5%) diabetes who were between the ages of 7-17 years of age. The purpose of the study was to determine the effect in glycemic control as measured by HgbA1c with use of iPro™ CGM at regularly scheduled clinic appointments. Recruitment for this study was limited to patients at the University of Texas Health Science Center in San Antonio Pediatric Diabetes Clinic from May 2011 to March 2013. Subjects were randomized into Group1 or Group 2 using sequentially numbered, opaque sealed envelopes (SNOSE).

All subjects had point-of-care HgbA1c (standard of care) and CGM data collected at time points 0, 3 months, and 6 months. After a regularly scheduled clinic appointment, all subjects and families at time 0 were counseled by a registered dietician regarding carbohydrate counting with a focus on minimizing errors in carbohydrate estimation, as is standard of care for patients with poorly controlled diabetes in our clinic. At time 0, subjects in both Group 1 and 2 had CGM placement after meeting with the dietician. Group 1 subjects were blinded to the first CGM data, meaning that they did not review the CGM download data. Group 2 was scheduled to return to clinic within 2 weeks of placement to meet with a pediatric endocrinologist involved in the study to interpret the CGM results and make adjustments to insulin regimen if appropriate. Both Groups 1 and 2 were not blinded to CGM data at 3 months and 6 months. Again, the CGM was placed after their regularly scheduled diabetes clinic appointments and all families returned within 2 weeks of these visits to meet with the pediatric endocrinologist to interpret the data and adjust the insulin regimen if necessary.

The iPro™ CGM was worn for a minimum of 48 hours (2 days), maximum 96 hours (4 days). Participants were instructed to complete a minimum of 4 SMBG records daily while wearing the iPro™ CGM for system calibration purposes. Subjects documented SMBGs, meal times, carbohydrate intake, insulin doses, exercise, and any hypoglycemic symptoms in a log book for correlation to CGM data.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of diabetes for at least 6 months, type 1 or type 2 diabetes.
2. Treated at UT Health Science Center pediatric diabetes clinic for at least the previous 3 months.
3. HgbA1c >8.5% (equivalent to average BG of >205 mg/dL for past three months).
4. Supportive family with willingness to self monitoring blood glucose values at least 4 times per day during study.
5. Supportive family with willingness to participate in continuous glucose monitoring (CGM) for at least 48 hours including self monitoring blood glucose values at least 4 times per day, documenting meals, carbohydrates eaten, insulin dose given, exercise, and hypoglycemic symptoms.
6. Attend proposed clinic, nutritional, and CGM follow up visits.
7. Pump or multiple daily injection (MDI) insulin therapy (3-4 injections minimum daily). If on pump, on pump for at least the past 3 months. Current insulin regimen involves basal/ bolus therapy with no plans to switch the modality of insulin administration during the study (e.g., injection user switching to a pump, pump user switching to injections).
8. Hypoglycemic unawareness.
9. English or Spanish primary language.

Exclusion Criteria:

1. Medications known to affect glycemic control (oral steroids, growth hormone, psychotropics).
2. Documented concomitant chronic disease known to affect glycemic control.
3. 3 or more incidents in the last 12 months of severe hypoglycemia with documented blood glucose below 50mg/dL (if possible), resulting in unconsciousness, hospitalization or third party assistance, where recovery follows treatment with glucose or glucagon or similar.
4. 3 or more incidents in the last 12 months of diabetic ketoacidosis (DKA).
5. Reported alcohol or drug abuse.
6. Documented cutaneous allergy to latex products.
7. Documented eating disorders or morbid obesity as assessed by the investigator.
8. Any other medical, social or psychological condition that, in the investigator's opinion, makes the patient unable to comply with the study protocol and all study procedures.
9. Home use of CGM in the past 6 months.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects are pediatric, with a clinical diagnosis of diabetes for at least 6 months, who have been treated in the diabetic clinic for at least 3 months previously.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rayas, MD, Principal Investigator — UT Health Science Center San Antonio

REFERENCES:
- [Background] Maahs DM, West NA, Lawrence JM, Mayer-Davis EJ. Epidemiology of type 1 diabetes. Endocrinol Metab Clin North Am. 2010 Sep;39(3):481-97. doi: 10.1016/j.ecl.2010.05.011. PMID 20723815
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Borus JS, Laffel L. Adherence challenges in the management of type 1 diabetes in adolescents: prevention and intervention. Curr Opin Pediatr. 2010 Aug;22(4):405-11. doi: 10.1097/MOP.0b013e32833a46a7. PMID 20489639
- [Background] Boland E, Monsod T, Delucia M, Brandt CA, Fernando S, Tamborlane WV. Limitations of conventional methods of self-monitoring of blood glucose: lessons learned from 3 days of continuous glucose sensing in pediatric patients with type 1 diabetes. Diabetes Care. 2001 Nov;24(11):1858-62. doi: 10.2337/diacare.24.11.1858. PMID 11679447
- [Background] Gandrud LM, Xing D, Kollman C, Block JM, Kunselman B, Wilson DM, Buckingham BA. The Medtronic Minimed Gold continuous glucose monitoring system: an effective means to discover hypo- and hyperglycemia in children under 7 years of age. Diabetes Technol Ther. 2007 Aug;9(4):307-16. doi: 10.1089/dia.2007.0026. PMID 17705686
- [Background] Bode BW, Gross TM, Thornton KR, Mastrototaro JJ. Continuous glucose monitoring used to adjust diabetes therapy improves glycosylated hemoglobin: a pilot study. Diabetes Res Clin Pract. 1999 Dec;46(3):183-90. doi: 10.1016/s0168-8227(99)00113-8. PMID 10624783
- [Background] Tanenberg R, Bode B, Lane W, Levetan C, Mestman J, Harmel AP, Tobian J, Gross T, Mastrototaro J. Use of the Continuous Glucose Monitoring System to guide therapy in patients with insulin-treated diabetes: a randomized controlled trial. Mayo Clin Proc. 2004 Dec;79(12):1521-6. doi: 10.4065/79.12.1521. PMID 15595336
- [Background] Chetty VT, Almulla A, Odueyungbo A, Thabane L. The effect of continuous subcutaneous glucose monitoring (CGMS) versus intermittent whole blood finger-stick glucose monitoring (SBGM) on hemoglobin A1c (HBA1c) levels in Type I diabetic patients: a systematic review. Diabetes Res Clin Pract. 2008 Jul;81(1):79-87. doi: 10.1016/j.diabres.2008.02.014. Epub 2008 Apr 15. PMID 18417243
- [Background] Kaufman FR, Gibson LC, Halvorson M, Carpenter S, Fisher LK, Pitukcheewanont P. A pilot study of the continuous glucose monitoring system: clinical decisions and glycemic control after its use in pediatric type 1 diabetic subjects. Diabetes Care. 2001 Dec;24(12):2030-4. doi: 10.2337/diacare.24.12.2030. PMID 11723078
- [Background] Ludvigsson J, Hanas R. Continuous subcutaneous glucose monitoring improved metabolic control in pediatric patients with type 1 diabetes: a controlled crossover study. Pediatrics. 2003 May;111(5 Pt 1):933-8. doi: 10.1542/peds.111.5.933. PMID 12728068
- [Background] Lagarde WH, Barrows FP, Davenport ML, Kang M, Guess HA, Calikoglu AS. Continuous subcutaneous glucose monitoring in children with type 1 diabetes mellitus: a single-blind, randomized, controlled trial. Pediatr Diabetes. 2006 Jun;7(3):159-64. doi: 10.1111/j.1399-543X.2006.00162.x. PMID 16787523
- [Background] Schaepelynck-Belicar P, Vague P, Simonin G, Lassmann-Vague V. Improved metabolic control in diabetic adolescents using the continuous glucose monitoring system (CGMS). Diabetes Metab. 2003 Dec;29(6):608-12. doi: 10.1016/s1262-3636(07)70076-9. PMID 14707890
- [Background] Ryan EA, Germsheid J. Use of continuous glucose monitoring system in the management of severe hypoglycemia. Diabetes Technol Ther. 2009 Oct;11(10):635-9. doi: 10.1089/dia.2009.0042. PMID 19821755
- [Result] Hood KK, Rohan JM, Peterson CM, Drotar D. Interventions with adherence-promoting components in pediatric type 1 diabetes: meta-analysis of their impact on glycemic control. Diabetes Care. 2010 Jul;33(7):1658-64. doi: 10.2337/dc09-2268. PMID 20587726
- [Result] Stanger C, Ryan SR, Delhey LM, Thrailkill K, Li Z, Li Z, Budney AJ. A multicomponent motivational intervention to improve adherence among adolescents with poorly controlled type 1 diabetes: a pilot study. J Pediatr Psychol. 2013 Jul;38(6):629-37. doi: 10.1093/jpepsy/jst032. Epub 2013 May 22. PMID 23699750
- [Result] Mulvaney SA, Hood KK, Schlundt DG, Osborn CY, Johnson KB, Rothman RL, Wallston KA. Development and initial validation of the barriers to diabetes adherence measure for adolescents. Diabetes Res Clin Pract. 2011 Oct;94(1):77-83. doi: 10.1016/j.diabres.2011.06.010. Epub 2011 Jul 7. PMID 21737172
- [Result] Telo GH, Volkening LK, Butler DA, Laffel LM. Salient characteristics of youth with type 1 diabetes initiating continuous glucose monitoring. Diabetes Technol Ther. 2015 Jun;17(6):373-8. doi: 10.1089/dia.2014.0290. Epub 2015 Mar 6. PMID 25749206

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Initially blinded to continuous glucose monitoring data
- Group 2: Never blinded to continuous glucose monitoring data
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 16 | 14
Completed | 10 | 9
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Initially blinded to continuous glucose monitoring data after 1st use Not blinded to continuous glucose monitoring data after 2nd and 3rd use
  continuous glucose monitoring (CGM): All subjects in Groups 1 and 2 wore the CGM device at time points 0, 3 months, and 6 months. Group 1 did not review CGM data at time 0, but did review CGM data at time point 3 months and 6 months. Group 2 reviewed CGM data at all time points.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (3.16) | 13 (3.05) | 12.74 (3.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Pubertal [Count of Participants; unit: Participants] | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Was Change in HgbA1c
Time Frame: 0 months, 3 months and 6 months
Measure: Median (Inter-Quartile Range); unit: HbgA1c %
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 10 | 9
HbgA1c %
  Change between 0 mo and 3 mo | -0.95 [-1.7 to 0.7] | -0.9 [-1.4 to -0.4]
  Change between 3 mo and 6 mo | -0.6 [-0.9 to -0.1] | -0.9 [-1.4 to -0.4]
  Change between 0 mo and 6 mo | -1.1 [-2.4 to 0] | -0.5 [-0.9 to 0.2]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Testing the change between two time points within each group using Wilcoxon signed rank test; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: % Time Spent in Hypoglycemia, Hyperglycemia, and Euglycemia
Time Frame: 3 months and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 3/16 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=16) | Group 2 (N=14)
Pain with catheter insertion (Skin and subcutaneous tissue disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No